CLINICAL TRIAL: NCT01049321
Title: The Effect of DASH Diet on the Cardiometabolic Risks and Hepatic Function Among Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Shahid Motahari Hospital of Fooladshahr, Isfahan Steel Company, Isfahan (Unknown)
Responsible Party: Isfahan University of medical sciences, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DASH and cardiovascular risks
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2008-03

CONDITIONS: Type 2 Diabetic Patients
Keywords: Dietary Approach to Stop Hypertension; weight; coagulation; DASH eating pattern.
MeSH Terms: conditions — Body Weight; Thrombosis | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DASH diet (Experimental): DASH: Dietary approaches to stop hypertension eating plan
  Interventions: Dietary Supplement: DASH diet
- Diabetic diet (Placebo Comparator): Diabetic diet: a usual diabetic diet
  Interventions: Dietary Supplement: a usual diabetic diet

INTERVENTIONS:
Dietary Supplement: DASH diet
  Other Names: Dietary aproaches to stop hypertension
  Arms: DASH diet
Dietary Supplement: a usual diabetic diet
  Arms: Diabetic diet

SUMMARY:
The investigators are not aware of any study regarding the effect of DASH eating pattern on different cardiovascular risks among type 2 diabetic patients. The investigators assumed that DASH eating pattern could reduce the cardio-metabolic risks and improve the hepatic function among type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Having type 2 diabetes

Exclusion Criteria:

* Having other chronic disease, hepatic or kidney disorders, cancer, hormone therapy

Ages: 44 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Cardio-metabolic risks | 6 months

SECONDARY OUTCOMES:
Hepatic function | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Leila Azadbakht, PhD, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Shahid motahari hospital, Esfahan Esteel company, Iran, Isfahan, Iran

REFERENCES:
- [Derived] Azadbakht L, Surkan PJ, Esmaillzadeh A, Willett WC. The Dietary Approaches to Stop Hypertension eating plan affects C-reactive protein, coagulation abnormalities, and hepatic function tests among type 2 diabetic patients. J Nutr. 2011 Jun;141(6):1083-8. doi: 10.3945/jn.110.136739. Epub 2011 Apr 27. PMID 21525259